CLINICAL TRIAL: NCT01171443
Title: Is There a Role of Oxidative Stress in the Pathophysiology of Bortezomib Induced Peripheral Neuropathy (BIPN) in Multiple Myeloma Patients?
Brief Title: The Pathophysiology of Bortezomib Induced Peripheral Neuropathy
Acronym: BIPN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dr' Ghoti Hossam, hematology department on Wolfsson Medical Center
Other Study IDs: 0102-10CTIL
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Since the pathophysiology of BIPN still remains unclear, in the present study we are going to assess the development of BIPN in newly diagnosed myeloma patients, based on clinical neurological examination and electrophysiological study (EMG) and trying to find out if there is any relationship between oxidative stress generation measured by serum malonyldialdehyde - (MDA) and urinary isoprostane, and the development of BIPN, which can explain important part of the BIPN pathophysiology and can suggest new ideas of treatment and prophylactic strategies of peripheral neuropathy.

DETAILED DESCRIPTION:
The proteasome inhibitor bortezomib has shown impressive clinical activity alone and in combination with other novel agents for the treatment of multiple myeloma (MM).

Peripheral neuropathy is a significant dose limiting toxicity of bortezomib, which typically occurs within the first treatment cycles with bortezomib, reaching plateau around cycle 5, and does not appear to increase thereafter.

Although bortezomib is known to be selective proteasome inhibitor, the mechanisms of cytotoxicity are poorly understood.

It has been theoretically hypothesized that bortezomib abrogates the degradation of I-kB, which blocks the transcriptional activity of NF-kB, however, recent studies demonstrated that bortezomib elicits activation of multiple pathways in cancer cells, such as reactive oxygen species (ROS) pathway.

The involvement of oxidative stress is supported by emerging studies showing that ROS generation plays a critical role in the initiation of the bortezomib induced apoptotic cascade.

Oxidative stress is a complex and dynamic situation characterized by an imbalance between the productions of ROS and the availability and action of antioxidants.

ELIGIBILITY:
Inclusion Criteria:

1. A total of 30 newly diagnosed patients (age > 18 years) with multiple myeloma (stage3 Durie and Salmon, ECOG-performance status <2), who are candidates for bortezomib therapy will be enrolled in the study (duration of the study 6 months).

Exclusion Criteria:

1. Patients with relapsed or progressive multiple myeloma.
2. Performance status > 2.
3. Prior treatment with neuropathic agents such as Oncovin and thalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 newly diagnosed patients (age > 18 years) with multiple myeloma (stage3 Durie and Salmon, ECOG-performance status <2), who are candidates for bortezomib therapy will be enrolled in the study (duration of the study 6 months).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GHOTI HOSSAM, Principal Investigator — HEMATOLOGY DEPARTMENT ON WOLFSSON MEDICAL CENTER
Locations (1):
- Wolfsson Medical Center, Holon, Israel, Israel